CLINICAL TRIAL: NCT00583544
Title: A Double Blind, Sequential, Ascending Single Dose, Placebo-Controlled Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Study of TC-2216 in Healthy Young Male Volunteers.
Brief Title: A Safety and Tolerability Single Ascending Dose Study in Healthy Volunteers
Acronym: SRD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Geoffrey Dunbar, Vice President, CDRA, Targacept, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-2216-232-CLP-001
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
Keywords: Healthy; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: TC-2216
- 2 (Experimental)
  Interventions: Drug: TC-2216

INTERVENTIONS:
Drug: TC-2216 — Multiple ascending dose groups will be explored.

SUMMARY:
Targacept, Inc. is studying TC-2216 for a potential role in the treatment of central nervous system (CNS) neurobiological disorders in anticipation of seeking an indication in depression and/or anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 18-40 years old (both ages included).
2. Subjects must be in good health as determined by their medical history, physical examination, psychological examination, ECG, vital signs, standard EEG and laboratory tests. A volunteer with a clinical abnormality may be included only if the Investigator or his designee considers that the abnormality will not introduce additional risk factor for the subject's health, or interfere with the study objectives.
3. Subjects with a body mass index within the range 18-29 kg/m2 and a weight within the range of 60-90 kg.
4. Non-smoker subjects (a cotinine test will be performed at screening and Day -1
5. Subjects must be able to refrain from consuming xanthine containing beverages, and must refrain from intensive physical exercise during the study conduct (until the end of study visit).
6. Subjects must have signed an informed consent form indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions.
7. Subjects must be affiliated with, or a beneficiary of, a French social security system.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Any clinically relevant acute or chronic diseases which could interfere with the subjects safety during the trial, or expose them to undue risk, or which could interfere with the study objectives.
2. History or presence of gastrointestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
3. Any history of drug or other significant allergy.
4. Likely to need any treatment (including dental care) during the study period.
5. Donation of one or more units of blood within 90 days prior to the screening.
6. Use of any prescription or over-the-counter medication within 14 days prior to admission on Day-1 (not including paracetamol in the range of 1gr/day). In addition any medications with central effects are prohibited for a period equal to 5 x half-life prior to admission (Day-1), should this period be longer than 14 days.
7. Alcohol consumption > 40 g alcohol/day (1 glass (25 cl) of beer with 3° of alcohol = 7.5 g, or 1 glass (25 cl) of beer with 6° of alcohol = 15 g, or 1 glass (12.5 cl) of wine with 10° of alcohol = 12 g, or 1 glass (4cl) of aperitif with 42° of alcohol = 17 g).
8. Positive alcotest at screening and Day -1 .
9. Positive test result on hepatitis B surface antigen, hepatitis C antibody.
10. Positive test result on HIV 1 and 2 serology.
11. Excessive daily consumption of xanthines containing drinks (i.e > 500 mg/day of caffeine).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
hematology, biochemistry, urine analysis, vital sign, ECG, adverse events. | 4 days

SECONDARY OUTCOMES:
plasma and urine pharmacokinetics, Pharmaco EEG, Bond-Lader Visual Analogue Scal | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Targacept Clinical Trials, MD, Study Director — Targacept Inc.
Locations (1):
- Forenap Pharma, Rouffache, France